CLINICAL TRIAL: NCT01278797
Title: A Single-Dose, Comparative Bioavailability Study of Telmisartan/Amlodipine 80 mg/10 mg Tablets Versus Micardis 80 mg Tablets With Norvasc 10 mg Tablets Under Fasting Conditions
Brief Title: Telmisartan and Amlodipine Versus Monocomponent Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1235.41
Record Dates: First submitted 2011-01-17; First posted 2011-01-19 (Estimated); Results first posted 2012-03-16 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — telmisartan amlodipine combination

ARMS (2):
- Telmisartan/Amlodipine Fixed Dose (Active Comparator): Telmisartan/Amlodipine medium fixed dose combination tablet once daily.
  Interventions: Drug: Telmisartan/Amlodipine Combination Tablet
- Amlodipine Monocomponent (Active Comparator): Amlodipine Monocomponent 10mg tablet once daily
  Interventions: Drug: Amlodipine Monocomponent

INTERVENTIONS:
Drug: Telmisartan/Amlodipine Combination Tablet — Combination Tablet
  Arms: Telmisartan/Amlodipine Fixed Dose
Drug: Amlodipine Monocomponent — Active Comparator
  Arms: Amlodipine Monocomponent

SUMMARY:
This study will be an open-label, randomized, two-treatment, two-period, two-sequence crossover study to evaluate the bioequivalence of the amlodipine component of Boehringer Ingelheim Pharma GmbH & Co. KGs 80 mg telmisartan/10 mg amlodipine fixed dose combination tablet to the corresponding mono-component amlodipine tablets, 10 mg (Pfizers Norvasc).

ELIGIBILITY:
Inclusion criteria:

1. Healthy, non-smoking, male and/or post-menopausal/surgically sterile female subjects from 18 to 55 years of age.
2. Females who participate in this study must either:

   1. be post-menopausal for at least 1 year (no menstrual cycle for 12 consecutive months) and deemed post-menopausal by a physician based on screening clinical laboratory tests (Follicle stimulating hormone (FSH) and Luteinising Hormone (LH)
   2. provide proof of surgical sterility.
3. Body Mass Index (BMI) greater than or equal to 19.0 and less than or equal to 30.0 kg/m2.
4. No clinically significant findings in vital signs measurements and systolic blood pressure greater than or equal to 110 mmHg at screening.
5. No clinically significant abnormal laboratory values.
6. No clinically significant findings in a 12-lead electrocardiogram (ECG) and the time between the P and the R waves on the ECG (PR interval) less than or equal to 200 ms at screening.
7. Have no significant diseases.
8. Be informed of the nature of the study and give written consent prior to receiving any study procedure.
9. Have no clinically significant findings from a physical examination.

Exclusion criteria:

1. Known history or presence of any clinically significant medical condition.
2. Known or suspected carcinoma.
3. History or presence of cardiovascular dysfunction (e.g. increased angina, myocardial infarction, outflow obstruction, congestive heart failure).
4. History of clinically significant hypotension.
5. Presence of hepatic dysfunction.
6. Known history or presence of galactose or fructose intolerance, sucrase-isomaltase insufficiency, Lapp lactase insufficiency, galactosemia, or glucose-galactose malabsorption syndrome.
7. History of gastrointestinal tract surgery (appendectomy is permitted).
8. Presence of clinically significant gastrointestinal disease or history of malabsorption within the last year.
9. Presence of a medical condition requiring regular medication (prescription and/or over-the-counter) with systemic absorption.
10. History of drug or alcohol addiction requiring treatment.
11. Positive test result for serum hCG consistent with pregnancy (females only), HIV, Hepatitis B surface antigen, or Hepatitis C antibody.
12. Positive test result for urine drugs of abuse (cannabinoids, opiates, amphetamines, cocaine, phencyclidine, tricyclic antidepressants, barbiturates, methadone, and benzodiazepines) or urine cotinine.
13. Difficulty fasting or consuming standard meals.
14. Females who are pregnant, lactating, or likely to become pregnant during the study.
15. Does not tolerate venipuncture.
16. Use of tobacco or nicotine-containing products within 6 months prior to drug administration.
17. On a special diet within 30 days prior to drug administration (e.g. liquid, protein, raw food diet).
18. Participated in another clinical trial or received an investigational product within 30 days prior to drug administration.
19. Donation or loss of whole blood:

    1. Great than or equal to 50 mL and less than or equal to 499 mL within 30 days prior to dosing
    2. greater than or equal to 500 mL within 56 days prior to dosing.
20. Females who have used hormonal contraceptives within 6 months prior to drug administration.
21. Have had a tattoo or body piercing within 30 days prior to dosing.
22. Known history or presence of hypersensitivity or idiosyncratic reaction to telmisartan, amlodipine, or any other drug substances with similar activity.
23. Use of any drugs known to:

    1. induce (e.g. barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole)
    2. inhibit (e.g. antidepressants (Selective Seratonin Reuptake Inhibitor (SSRI)I), cimetidine, diltiazem, macrolides, imidazoles, neuroleptics, verapamil, fluoroquinolones, antihistamines) hepatic drug metabolism within 30 days prior to drug administration.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2011-01; Primary Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1235.41.0001 Boehringer Ingelheim Investigational Site, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Telm/Amlo 80 mg/10 mg First, Then Telm 80 mg + Amlo 10 mg: Combination tablet followed by individual components
- Telm 80 mg + Amlo 10 mg First, Then Telm/Amlo 80 mg/10 mg: Individual components followed by Combination tablet
Period: Period 1
Arm/Group | Telm/Amlo 80 mg/10 mg First, Then Telm 80 mg + Amlo 10 mg | Telm 80 mg + Amlo 10 mg First, Then Telm/Amlo 80 mg/10 mg
Started | 14 | 14
Completed | 13 | 13
Not Completed | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 1 | 0
Period: Washout Period of 21 Days
Arm/Group | Telm/Amlo 80 mg/10 mg First, Then Telm 80 mg + Amlo 10 mg | Telm 80 mg + Amlo 10 mg First, Then Telm/Amlo 80 mg/10 mg
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Telm/Amlo 80 mg/10 mg First, Then Telm 80 mg + Amlo 10 mg | Telm 80 mg + Amlo 10 mg First, Then Telm/Amlo 80 mg/10 mg
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes all subjects randomized to either treatment sequence
Arm/Group | Entire Study Population
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 27
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic/Latino | 7
  Asian | 3
  Black/African American | 6
  White | 12
Height [Mean (Standard Deviation); unit: centimeter] | 173.1 (7.1)
Weight [Mean (Standard Deviation); unit: kilogram] | 80.3 (9.9)
Body Mass Index [Mean (Standard Deviation); unit: kilogram / square meter] | 26.7 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of Plasma Amlodipine From 0 to 72 Hours (AUC72)
Description: Area under the analyte concentration versus time curve from time zero to 72 hours as calculated by the linear trapezoidal method
Time Frame: Day 1, Day 22
Population: Analysis Set includes all randomized participants who completed the trial
Measure: Mean (Standard Deviation); unit: nanograms*hour/milliliter
Groups:
- Telm/Amlo 80 mg/10 mg: Combination tablet
- Telm 80 mg + Amlo 10 mg: Individual tablets
Arm/Group | Telm/Amlo 80 mg/10 mg | Telm 80 mg + Amlo 10 mg
Number analyzed (Participants) | 26 | 26
nanograms*hour/milliliter | 260.7971 (60.8717) | 276.6315 (66.1935)
Statistical Analysis 1: Comparison: Telm/Amlo 80 mg/10 mg vs Telm 80 mg + Amlo 10 mg; Telmisartan/Amlodipine 80 mg/10 mg versus Telmisartan 80 mg + Amlodipine 10 mg The two formulations are shown to be bioequivalent since the 90% confidence interval of the test to reference ratio is entirely contained within the 80-125% bioequivalence range; Test type: Superiority or Other; p = 0.005, ANOVA; ANOVA was applied to log-transformed AUC72 and Included treatment, sequence, period and subject-within-sequence effects; Test/Reference ratio of geometric means = 94.51, 90% CI [91.60 to 97.51]

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Amlodipine
Time Frame: Day 1, Day 22
Population: Analysis Set includes all randomized participants who completed the trial
Measure: Mean (Standard Deviation); unit: nanograms/milliliter
Arm/Group | Telm/Amlo 80 mg/10 mg | Telm 80 mg + Amlo 10 mg
Number analyzed (Participants) | 26 | 26
nanograms/milliliter | 6.7465 (1.3354) | 7.2258 (1.6549)
Statistical Analysis 1: Comparison: Telm/Amlo 80 mg/10 mg vs Telm 80 mg + Amlo 10 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0093, ANOVA; ANOVA was applied to log-transformed CMAX and Included treatment, sequence, period and subject-within-sequence effects; Test/Reference ratio of geometric means = 94.10, 90% CI [90.70 to 97.63]

3. Secondary Outcome: Time of Maximum Concentration of Amlodipine (TMAX)
Description: Time of maximum measured amlodipine concentration over the zero to 72 hour sampling period
Time Frame: Day 1, Day 22
Population: Analysis Set includes all randomized participants who completed the trial
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Telm/Amlo 80 mg/10 mg | Telm 80 mg + Amlo 10 mg
Number analyzed (Participants) | 26 | 26
hours | 6.69 (1.95) | 6.12 (1.40)
Statistical Analysis 1: Comparison: Telm/Amlo 80 mg/10 mg vs Telm 80 mg + Amlo 10 mg; Telmisartan/Amlodipine 80 mg/10 mg versus Telmisartan 80 mg + Amlodipine 10 mg; Test type: Superiority or Other; p = 0.153, ANOVA; ANOVA was applied to TMAX and Included treatment, sequence, period and subject-within-sequence effects; Mean Difference (Final Values) = 0.58

ADVERSE EVENTS:
Time Frame: 30 Days
Arm/Group | Telm/Amlo 80 mg/10 mg | Telm 80 mg + Amlo 10 mg
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 3/27 | 3/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Telm/Amlo 80 mg/10 mg (N=27) | Telm 80 mg + Amlo 10 mg (N=27)
Blood urine present (Renal and urinary disorders) | 1 | 2
Headache (Nervous system disorders) | 2 | 1
Urine abnormality (Renal and urinary disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.